CLINICAL TRIAL: NCT03884439
Title: Infliximab BS for Intravenous Drip Infusion 100 mg "Pfizer" General Investigation (Crohn's Disease or Ulcerative Colitis)
Brief Title: Infliximab Biosimilar "Pfizer" Drug Use Investigation (Crohn's Disease or Ulcerative Colitis)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B5371008
Record Dates: First submitted 2019-03-04; First posted 2019-03-21 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's Disease; Ulcerative Colitis; Infliximab; biosimilar
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab [infliximab biosimilar 3]: Patients with Crohn's Disease or Ulcerative Colitis treated by Infliximab BS
  Interventions: Drug: Infliximab [infliximab biosimilar 3]

INTERVENTIONS:
Drug: Infliximab [infliximab biosimilar 3] — <Crohn's disease> The usual dose is 5 mg as Infliximab [Infliximab Biosimilar 3] for every kg of body weight given as an intravenous infusion. After an initial dose is given, the subsequent doses are given at Weeks 2 and 6, and every 8 weeks thereafter. After a dose at Week 6 is given, the dose may be increased or the dosing interval may be reduced for patients who have reduced effects. At an increased dose, the dose may be adjusted to 10 mg for every kg of body weight. At a reduced dosing interval, the dose of 5 mg for every kg of body weight may be given at the minimum dosing interval of 4 weeks. <Ulcerative colitis> The usual dose is 5 mg as Infliximab [Infliximab Biosimilar 3] for every kg of body weight given as an intravenous infusion. After an initial dose is given, the subsequent doses are given at Weeks 2 and 6, and every 8 weeks thereafter.
  Other Names: Infliximab BS for Intravenous Drip Infusion 100 mg "Pfizer"

SUMMARY:
To collect information on the safety and effectiveness of Infliximab BS for Intravenous Drip Infusion 100 mg "Pfizer" against Crohn's disease or ulcerative colitis under actual status of use.

DETAILED DESCRIPTION:
This study will be conducted with all-case investigation system in patients with Crohn's disease or ulcerative colitis.

This study will be conducted in patients who used this drug after the day of approval of dosage and administration for Crohn's disease or ulcerative colitis at contracted medical institutions. Patients who used this drug before conclusion of the contract with the medical institution will also be included in this study (retrospective patients will be included).

Therefore, Time Perspective is retrospective and prospective.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease or ulcerative colitis who started treatment with this drug
* Patients who received this drug for the first time at the medical institution after the day of launch of this drug.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Crohn's Disease or Ulcerative Colitis treated by Infliximab BS
Sampling Method: Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local Country Office, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5371008

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]: Participants with Crohn's disease or Ulcerative colitis who received Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] as indicated in the approved local product document for the first time were observed for 30 weeks from the day of initial dose of this drug. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Started | 416
Completed | 371
Not Completed | 45
Not completed — No informed consent for publication of study results | 38
Not completed — Contract violation/deficiency | 7

BASELINE CHARACTERISTICS:
Population: A total of 416 participants started the study. Of the 416 participants, 371 completed the study.
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 371
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 353
  ≥65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 271
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was a treatment-related adverse event, and any untoward medical occurrence attributed to Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] in a participant who received this drug. Relatedness to Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] was assessed by the physician.
Time Frame: 30 weeks from the day of initial dose
Population: The safety analysis set (371 participants) comprised of participants who satisfied the inclusion criteria and had received Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]. Participants with no informed consent for publication of study results and contract violation/deficiency were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 371
Participants | 7

2. Secondary Outcome: Percentage of Participants With Remission (Crohn's Disease Activity Index [CDAI]) for Crohn's Disease
Description: Percentage of participants with remission of Crohn's disease was presented using the Crohn's Disease Activity Index score along with the two-sided 95% confidence interval (exact method).
  The Crohn's Disease Activity Index score is calculated from the following 8 items: (1) the number of watery or mushy stools, (2) abdominal pain (0 to 3), (3) general condition (0 to 4), (4) symptoms and signs considered to be related to Crohn's disease (0 to6), (5) use of Lomotil/Opiate for diarrhea (0 to 1), (6) abdominal mass (0 to 5), (7) hematocrit(%), and (8) score derived from body weight, that is the sum of 2x(1)+5x(2)+7x(3)+20x(4)+30x(5)+10x(6)+6x(7)+(8). A Crohn's Disease Activity IndexI score of <150 was considered remission.
Time Frame: Baseline, Study comnletion date which is the day of visit immediately after 8 weeks have elapsed since the last dose during the observation period.
Population: The efficacy analysis set (348 participants) comprised of participants in the safety analysis set who had effectiveness evaluation. Of the 348 participants, percentage of remission and improvement of Crohn's disease as of the end date of the study was calculated for the 151 participants whose effectiveness was evaluated by the CDAI score.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 151
Percentage of participants
  At baseline | 84.1 [77.28 to 89.54]
  At study completion date | 87.4 [81.05 to 92.25]

3. Secondary Outcome: Percentage of Participants With Improvement the Crohn's Disease Activity Index for Crohn's Disease
Description: Percentage of participants with improvement of Crohn's disease was presented using the Crohn's Disease Activity Index score along with the two-sided 95% confidence interval (exact method).
  The Crohn's Disease Activity Index score is calculated from the following 8 items:(1) the number of watery or mushy stools, (2) abdominal pain (0 to 3), (3) general condition (0 to 4), (4) symptoms and signs considered to be related to Crohn's disease (0 to6), (5) use of Lomotil/Opiate for diarrhea (0 to 1), (6) abdominal mass (0 to 5), (7) hematocrit(%), and (8) score derived from body weight, that is the sum of 2x(1)+5x(2)+7x(3)+20x(4)+30x(5)+10x(6)+6x(7)+(8). The Crohn's Disease Activity Index improvement was defined as a decrease of 25% or more and 70 points or more in Crohn's Disease Activity Index score after treatment with Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] compared with the Crohn's Disease Activity Index score before treatment.
Time Frame: Study comnletion date which is the day of visit immediately after 8 weeks have elapsed since the last dose during the observation period.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 151
Percentage of participants | 6.6 [3.22 to 11.84]

4. Secondary Outcome: Percentage of Participants With Remission (Partial Mayo) Score for Ulcerative Colitis
Description: Percentage of participants with remission of Ulcerative colitis was presented using the partial Mayo score along with the two-sided 95% confidence interval (exact method).
  The partial Mayo score is the sum of the subscores for the following 3 domains with a range of 0 to 9 points; the number of bowel movements subscore (0 to 3), rectal bleeding subscore (0 to 3), and physician's global assessment subscore (0 to 3). Partial Mayo score of <2 was considered partial Mayo score remission.
Time Frame: as for outcome 2
Population: The efficacy analysis set (348 participants) comprised of participants in the safety analysis set who had effectiveness evaluation. Of the 348 participants, percentage of remission and improvement of Ulcerative colitis as of the end date of the study was calculated for the 87 participants whose effectiveness was evaluated by the partial Mayo score.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 87
Percentage of participants
  At baseline | 43.7 [33.06 to 54.74]
  At study completion date | 59.8 [48.71 to 70.15]

5. Secondary Outcome: Percentage of Participants With Improvement (Partial Mayo) Score for Ulcerative Colitis
Description: Percentage of participants with improvement of Ulcerative colitis was presented using the partial Mayo score along with the two-sided 95% confidence interval (exact method).
  The partial Mayo score is the sum of the subscores for the following 3 domains with a range of 0 to 9 points; the number of bowel movements subscore (0 to 3), rectal bleeding subscore (0 to 3), and physician's global assessment subscore (0 to 3). Partial Mayo score improvement was defined as 2 points or more reduction from baseline.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 87
Percentage of participants | 34.5 [24.61 to 45.44]

6. Secondary Outcome: Change of Mayo Score From Baseline to Study Completion Date for Ulcerative Colitis
Description: Summary statistics of the Mayo score at baseline, at study completion date, and the change in Mayo score from baseline to study completion date in participants with Ulcerative colitis.
  The Mayo score consists of 4 domains, each scored as a 0- to 3-point subscore, with higher scores indicating more severe disease activity. The 4 domains are the number of bowel movements subscore (0 to 3), rectal bleeding subscore (0 to 3), endoscopic finding subscore (0 to 3), and physician's global assessment subscore (0 to 3). The method of calculating the Mayo score is the sum of all subscores in the 4 domains, with a range of 0 to 12 points.
Time Frame: as for outcome 2
Population: The efficacy analysis set (348 participants) comprised of participants in the safety analysis set who had effectiveness evaluation. Of the 348 participants, summary statistics and change of the Mayo score was calculated for the 15 participants with Ulcerative colitis whose effectiveness was evaluated by the Mayo score.
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 15
Points on a scale
  At baseline | 5.0 (3.7)
  At study completion date | 3.1 (3.5)
  Change | -1.9 (2.7)

ADVERSE EVENTS:
Time Frame: 30 weeks from the day of initial dose
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
All-Cause Mortality (participants affected / at risk) | 0/371
Serious Adverse Events (participants affected / at risk) | 3/371
Other Adverse Events (participants affected / at risk) | 12/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] (N=371)
Cholelithiasis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] (N=371)
Tachycardia (Cardiac disorders) | 1
Auricular swelling (Ear and labyrinth disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Intestinal stenosis (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT03884439/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT03884439/SAP_001.pdf